CLINICAL TRIAL: NCT00576186
Title: Validation of the Gated Blood Pool SPECT: Comparison to ERNA and 3-dimensional Echocardiography.
Brief Title: Validation of the Gated Blood Pool SPECT: ERNA vs 3D Echo
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 27168
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Congestive Heart Failure; Ventricular Function, Left
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients being referred for the routine Equilibrium Radionuclide Angiocardiography (ERNA) for assessment of their left ventricular function will be asked to participate in the study. All patients will be asked to sign the consent form. Patients will be given a choice to participate in either or both studies (i.e. ERNA plus ACGBS or ERNA plus ACGBS and 3 DE).

SUMMARY:
This research study is designed to evaluate the accuracy of the techniques that are used to analyze heart function. The main purpose of this study is to analyze and compare three different methods of assessment of regional and overall heart function.

DETAILED DESCRIPTION:
The purpose of the present study is to establish the reproducibility and to validate gated blood pool SPECT imaging with application of attenuation correction (ACGBS) in evaluation of left ventricular regional and global function and volumes, by direct comparison with Equilibrium Radionuclide Angiocardiography (ERNA) and 3-dimensional ECHO (3DE).

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for routine clinically requested ERNA study for ejection fraction measurement at the Yale University Cardiovascular Nuclear Imaging Laboratory are eligible to be enrolled in the study.

Exclusion Criteria:

* Unstable medical condition preventing additional imaging.
* Weight greater than 300lbs, prohibiting imaging on the SPECT/CT imaging system.
* Patients with intracardiac shunts, emphysema or previously demonstrated allergies to octafluoropropane (the gas in the microbubbles), will not receive intravenous contrast during 3 DE image acquisition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient scheduled to undergo clinically requested ERNA imaging for assessment of LV function in the Yale University Cardiovascular Nuclear Imaging Laboratory will be an eligible candidate and will be asked to participate. Based on our referral pattern it will include both patients with cardiac and non-cardiac disease, the later usually consist of patients undergoing chemotherapy.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
2D echo provides a good estimate of regional LV function but if done with 3D analysis can provide a good estimate of global LV function and volumes. The quality of 3DE can be further improved by use of IV contrast which is FDA approved. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Sinusas, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Daou D, Coaguila C, Benada A, Razzouk M, Haidar M, Colin P, Lebtahi R, Slama M, Guludec DL. The value of a completely automatic ECG gated blood pool SPECT processing method for the estimation of global systolic left ventricular function. Nucl Med Commun. 2004 Mar;25(3):271-6. doi: 10.1097/00006231-200403000-00010. PMID 15094446
- [Background] Slart RH, Poot L, Piers DA, van Veldhuisen DJ, Nichols K, Jager PL. Gated blood-pool SPECT automated versus manual left ventricular function calculations. Nucl Med Commun. 2004 Jan;25(1):75-80. doi: 10.1097/00006231-200401000-00011. PMID 15061268
- [Background] De Bondt P, Nichols K, Vandenberghe S, Segers P, De Winter O, Van de Wiele C, Verdonck P, Shazad A, Shoyeb AH, De Sutter J. Validation of gated blood-pool SPECT cardiac measurements tested using a biventricular dynamic physical phantom. J Nucl Med. 2003 Jun;44(6):967-72. PMID 12791827
- [Background] Groch MW, DePuey EG, Belzberg AC, Erwin WD, Kamran M, Barnett CA, Hendel RC, Spies SM, Ali A, Marshall RC. Planar imaging versus gated blood-pool SPECT for the assessment of ventricular performance: a multicenter study. J Nucl Med. 2001 Dec;42(12):1773-9. PMID 11752072
- [Background] Mondelli JA, Di Luzio S, Nagaraj A, Kane BJ, Smulevitz B, Nagaraj AV, Greene R, McPherson DD, Rigolin VH. The validation of volumetric real-time 3-dimensional echocardiography for the determination of left ventricular function. J Am Soc Echocardiogr. 2001 Oct;14(10):994-1000. doi: 10.1067/mje.2001.115770. PMID 11593204
- [Background] Nosir YF, Salustri A, Kasprzak JD, Breburda CS, Ten Cate FJ, Roelandt JR. Left ventricular ejection fraction in patients with normal and distorted left ventricular shape by three-dimensional echocardiographic methods: a comparison with radionuclide angiography. J Am Soc Echocardiogr. 1998 Jun;11(6):620-30. doi: 10.1016/s0894-7317(98)70038-0. PMID 9657401
- [Background] Kuhl HP, Schreckenberg M, Rulands D, Katoh M, Schafer W, Schummers G, Bucker A, Hanrath P, Franke A. High-resolution transthoracic real-time three-dimensional echocardiography: quantitation of cardiac volumes and function using semi-automatic border detection and comparison with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Jun 2;43(11):2083-90. doi: 10.1016/j.jacc.2004.01.037. PMID 15172417
- [Background] Lee D, Fuisz AR, Fan PH, Hsu TL, Liu CP, Chiang HT. Real-time 3-dimensional echocardiographic evaluation of left ventricular volume: correlation with magnetic resonance imaging--a validation study. J Am Soc Echocardiogr. 2001 Oct;14(10):1001-9. doi: 10.1067/mje.2001.113647. PMID 11593205